CLINICAL TRIAL: NCT06913894
Title: Supervised Therapy Versus a Standardized Home-Based Program Versus No Formal Therapy for Uncomplicated, Nonoperatively Treated Distal Radius Fracture in Adults Under 50: A Three-Arm, Parallel-Group Randomized Controlled Trial
Brief Title: Supervised vs. Home-Based vs. No Therapy for Uncomplicated Distal Radius Fracture in Younger Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Al Hayah University In Cairo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DRFRecov2025-01
Record Dates: First submitted 2025-03-31; First posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-03

CONDITIONS: Distal Radius Fractures
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Intervention Model Description: Eligible adults will be randomly assigned to one of three groups: Supervised Therapy, Home-Based Program, or No Therapy. The groups differ only in the rehabilitation method post-cast removal, with all participants followed for 6 months.
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Supervised Therapy Group (STG) (Experimental): Participants will attend once-weekly supervised outpatient sessions (30-45 min) with a physical therapist for 6 weeks, in addition to a daily home exercise program (10-15 min).
  Interventions: Behavioral: Supervised Therapy for DRF Rehabilitation
- Home-Based Program Group (HBG) (Experimental): Participants perform a standardized home exercise program daily with weekly telephone or video follow-up (10 min sessions) over 6 weeks.
  Interventions: Behavioral: Home-Based Rehabilitation Program for DRF
- No Therapy Group (NTG) (Active Comparator): Participants receive minimal instruction via a general educational brochure (e.g., "move your wrist as tolerated") without formal exercise supervision.
  Interventions: Behavioral: Minimal Educational Intervention for DRF

INTERVENTIONS:
Behavioral: Supervised Therapy for DRF Rehabilitation — Participants assigned to the Supervised Therapy Group (STG) will receive in-person, supervised rehabilitation sessions in an outpatient clinic. Each session lasts 30-45 minutes and is conducted by a licensed physical therapist. The therapy focuses on progressive range of motion exercises, light strengthening, proprioception training, and functional task practice. In addition, participants are prescribed a daily home exercise program (lasting 10-15 minutes) to reinforce gains made during the clinic sessions. The intervention is provided over a 6-week period following cast removal, with adherence monitored via attendance records and home exercise logs.
  Arms: Supervised Therapy Group (STG)
Behavioral: Home-Based Rehabilitation Program for DRF — Participants assigned to the Home-Based Program Group (HBG) will follow a standardized, detailed home exercise program specifically designed for distal radius fracture rehabilitation. The program includes instructions for range of motion, strengthening, and functional tasks similar to the supervised protocol. Participants receive a comprehensive written and online exercise manual, and they are instructed to perform the exercises daily. In addition, they will have weekly telephone or video check-ins (approximately 10 minutes per call) with a research assistant to review progress, address questions, and ensure proper exercise technique. The home program is implemented over a 6-week period following cast removal, with adherence documented via exercise logs submitted by participants.
  Arms: Home-Based Program Group (HBG)
Behavioral: Minimal Educational Intervention for DRF — Participants assigned to the No Therapy Group (NTG) will receive a minimal intervention consisting solely of general educational material. At the time of cast removal, they will be provided with a simple, standardized educational brochure that contains basic instructions for wrist and hand movement (e.g., "move your wrist as tolerated"). No additional therapy sessions, home exercise logs, or follow-up telephone calls will be provided beyond routine care. This intervention is intended to reflect the absence of a formal rehabilitation program and serves as the control for evaluating the added benefit of supervised and home-based therapy.
  Arms: No Therapy Group (NTG)

SUMMARY:
This three-arm, parallel-group RCT will compare the effectiveness of three rehabilitation strategies following conservative treatment of an uncomplicated distal radius fracture in adults under 50 years old. The study will compare:

Supervised Therapy: Outpatient physical therapy sessions plus a daily home exercise program Home-Based Program: A structured, detailed home exercise program with weekly telephone follow-up No Therapy (minimal intervention): Standard minimal instruction via an educational brochure The primary outcome is the Patient-Rated Wrist Evaluation (PRWE) measured at 6 weeks and 6 months.

DETAILED DESCRIPTION:
Uncomplicated, nonoperatively treated distal radius fractures in younger adults (18-50 years) are common, yet current guidelines offer a "D" rating regarding optimal rehabilitation-specifically, whether structured, supervised therapy, a detailed home-based program, or no formal therapy is best. A lack of consensus may delay optimal recovery and unnecessarily increase healthcare usage.

After cast removal (typically 4-6 weeks), eligible participants will be randomized into one of three groups:

Supervised Therapy Group (STG): Participants attend once-weekly, 30- to 45-minute outpatient sessions with a licensed physical therapist for 6 weeks, focusing on progressive range of motion, light strengthening, proprioception, and functional tasks. They also perform a short daily home exercise program (10-15 minutes).

Home-Based Program Group (HBG): Participants perform a standardized, detailed exercise program at home, self-administered daily. They receive weekly phone or video follow-up (approximately 10 minutes) from research assistants.

No Therapy Group (NTG): Participants receive minimal instructions and an educational brochure (e.g., "move your wrist as tolerated") without formal exercise supervision.

Intervention components follow the TIDieR (Template for Intervention Description and Replication) guidelines:

Materials:

STG: Standard therapy equipment (theraband, therapy putty). HBG: Written and online exercise manual; exercise logs for self-report. NTG: General educational brochure.

Procedures:

STG: In-person 30-45-minute sessions weekly, plus daily home exercises. HBG: Self-directed exercise program with weekly telephonic check-ins. NTG: Minimal instruction only.

Who Provides:

STG: Licensed physical therapists. HBG: Research assistants provide check-ins. NTG: No active provider contact.

Where:

STG: Outpatient clinic visits. HBG: Participant's home with telephone support. NTG: No additional intervention setting.

When and How Much:

Duration: 6 weeks of intervention post-cast removal; full study follow-up over 6 months.

Frequency: STG = 1 clinical session per week + daily (~10-15 minute) home exercises; HBG = daily home routine with 1 weekly call; NTG = educational brochure at baseline.

Modifications:

Adjust therapy intensity for pain or reported complications; referral back to the treating surgeon if necessary.

Adherence:

STG attendance is tracked; HBG requires exercise logs; NTG has no structured adherence measures.

Planned Assessments:

Baseline (at cast removal), 6 weeks, 3 months, and 6 months follow-up.

ELIGIBILITY:
Inclusion Criteria:

Adults aged 18-50 years. Diagnosed with an extra-articular, stable distal radius fracture treated nonoperatively with a short-arm cast for approximately 4-6 weeks.

The fracture is uncomplicated (no significant soft-tissue injury, no evidence of CRPS, and no other major complications).

Willing to provide written informed consent and comply with follow-up assessments.

Exclusion Criteria:

Intra-articular or unstable fracture patterns. Surgical intervention planned or performed for the distal radius fracture. Presence of significant comorbidities (e.g., chronic inflammatory arthritis or severe neurological impairment affecting the injured limb).

Fracture complications such as CRPS or major soft-tissue injury. Inability to comply with study procedures or follow-up assessments. Pregnant or breastfeeding individuals.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2025-04-21 (Estimated); Primary Completion 2026-04-21 (Estimated); Study Completion 2026-04-21 (Estimated)

PRIMARY OUTCOMES:
Patient-Rated Wrist Evaluation (PRWE) Total Score | Assessed at 6 weeks (Cast-removal), 3 months, and 6 months post-intervention.
  The PRWE is a validated instrument assessing wrist pain and disability on a 0-100 scale (lower scores indicate better outcomes).

SECONDARY OUTCOMES:
Wrist/Forearm Range of Motion (ROM) | Assessed at 6 weeks (Cast-removal), 3 months, and 6 months post-intervention.
  ROM will be measured using a standard goniometer.
Upper Limb Disability (QuickDASH) | Assessed at 6 weeks (Cast-removal), 3 months, and 6 months post-intervention.
  The QuickDASH is an 11-item questionnaire evaluating upper limb function; lower scores indicate less disability.
Return-to-Activity Timeline | Recorded at 3 and 6 months post-intervention.
  The number of days required to resume work and/or sports will be documented.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy, Al Hayah University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No